CLINICAL TRIAL: NCT06229366
Title: [Ac-225]-PSMA-62 Phase I/II Clinical Trial to Characterize Efficacy, Safety, Tolerability, and Dosimetry in Oligometastatic Hormone Sensitive and Metastatic Castration Resistant Prostate Cancer (ACCEL)
Brief Title: [Ac-225]-PSMA-62 Trial in Oligometastatic Hormone Sensitive and Metastatic Castration Resistant Prostate Cancer
Acronym: ACCEL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27197; J5N-OX-JJEA (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-01-03; First posted 2024-01-29 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Metastatic Castration-resistant Prostate Cancer; Oligometastatic Prostate Carcinoma; Hormone Sensitive Prostate Cancer
Keywords: mCRPC; OmHSPC; Prostatic Neoplasms; Genital Neoplasms, Male; Castration Resistant Prostate Cancer; Hormone Sensitive Prostate Cancer; Oligometastatic Prostate Cancer; [225Ac]-PSMA-62; Ac-225-PSMA-62; Actinium; Radioligand Therapy; Radiopharmaceuticals; Urogenital Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OmHSPC (Experimental): Patients with prostate cancer and biochemical recurrence after definitive surgery or radiation therapy, with 1-5 PSMA-positive lesions, who have not yet initiated lifelong hormone therapy.
  Interventions: Drug: [Ac-225]-PSMA-62 (OmHSPC)
- mCRPC (Experimental): Patients with PSMA-positive mCRPC who have prior treatment with at least one APRI and received taxane chemotherapy (or ineligible/refused); and received a maximum of 3 prior systemic therapy regimens in the mCRPC setting.
  Interventions: Drug: [Ac-225]-PSMA-62 (mCRPC)

INTERVENTIONS:
Drug: [Ac-225]-PSMA-62 (mCRPC) — Phase Ia: Administered intravenously per dose escalation scheme. Patients will receive a single dose of [Ac-225]-PSMA-62 on Day 1 of each 6-week cycle for up to 4 cycles.
  Phase Ib: Administered intravenously at MTD or one dose level below MTD. Patients will receive a single dose of [Ac-225]-PSMA-62 on Day 1 of each 6-week or 4-week cycle, for a total of 4 cycles.
  Arms: mCRPC
Drug: [Ac-225]-PSMA-62 (OmHSPC) — Phase Ia: Administered intravenously per dose escalation scheme. Patients will receive a single dose of [Ac-225]-PSMA-62 on Day 1 of each 8-week cycle for up to 2 cycles.
  Phase Ib: Administered intravenously at MTD or one dose level below MTD. Patients will receive a single dose of [Ac-225]-PSMA-62 on Day 1 of each 8-week cycle, for a total of 2 cycles.
  Arms: OmHSPC

SUMMARY:
ACCEL is a multicenter, open label phase Ia/Ib/II study of [Ac-225]-PSMA-62 in participants with prostate-specific membrane antigen (PSMA)-positive prostate cancer.

DETAILED DESCRIPTION:
The primary aim of the phase Ia study is to evaluate the safety and tolerability of [Ac-225]-PSMA-62 to determine the maximum tolerated dose (MTD). The primary aim of the randomized phase Ib dose optimization is to determine the recommended phase II doses (RP2D) for patients with mCRPC and OmHSPC. The aim of the phase II study for patients with mCRPC is to evaluate the efficacy of [Ac-225]-PSMA-62.

ELIGIBILITY:
Inclusion Criteria:

1. Histological, pathological, and/or cytological confirmation of adenocarcinoma of the prostate
2. ECOG performance status 0 to 1
3. Criteria specific for patients with mCRPC:

   1. Previously received an androgen receptor pathway inhibitor (ARPI) and taxane-based chemotherapy (unless ineligible or refused taxane). Received a maximum of 3 prior systemic therapy regimens in the mCRPC setting
   2. Progressive mCRPC at the time of consent based on at least 1 of the following criteria being met in the context of castrate levels of testosterone:

      * PSA progression defined as rising PSA values at a minimum of 1-week intervals, with the last result being at least 1.0 ng/mL
      * Soft-tissue progression defined as an increase ≥20% in the sum of the diameter (SOD) (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD since treatment started or the appearance of one or more new lesions
      * Progression of bone disease defined as the appearance of two or more new lesions by bone scan
   3. At least one PSMA-PET positive lesion for prostate cancer
   4. Castrate circulating testosterone levels (<1.74 nmol/L or <50 ng/dL)
4. Criteria specific for patients with OmHSPC:

   1. PSA recurrence after radical prostatectomy (RP) or definitive radiation therapy (RT), with or without adjuvant/salvage local therapy (radiation or surgery), with or without (neo)adjuvant ADT

      * PSA ≥ 0.2ng/mL for patients with prior RP +/- RT, or
      * PSA of ≥ 2 ng/mL above nadir for patients with only prior RT
   2. 1- 5 PSMA-PET positive lesions identified outside the prostate bed or remaining gland.

Exclusion Criteria:

1. Patient has received any other investigational therapeutic agents within 4 weeks or 5 half-lives (whichever is shorter) of starting the study treatment
2. Evidence of ongoing and untreated urinary tract obstruction
3. Existing Grade 1 dry mouth (xerostomia) or symptomatic Grade 1 dry eye (xerophthalmia) for any reason
4. Patient has any concurrent severe and/or uncontrolled medical conditions that could increase the patient's risk for toxicity while on the study or that could confound discrimination between disease- and study treatment-related toxicities
5. Criteria specific for patients with mCRPC:

   1. Patient has received any PSMA-directed radioligand therapy (e.g., Lu-177-PSMA, Lu-177-PNT2002, Ac-225-J591)
   2. Patient has received any therapeutic systemic radionuclides (e.g., radium-223, rhenium-186, strontium-89), or non-PSMA-directed therapeutic radioligands (e.g., Lu-177-Dotatate) within 5 half-lives of starting the study treatment
6. Criteria specific for patients with OmHSPC:

   1. Patient has received any systemic anti-cancer therapy for prostate cancer with the exception of (neo)adjuvant ADT for management of localized disease
   2. Presence of any liver metastases
   3. Known presence of central nervous system metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | From first dose of study drug through end of DLT period (4 weeks)
  Phase Ia: Incidence of dose limiting toxicities (DLTs)
Safety, tolerability, and Recommended Phase II Dose (RP2D) | From first dose of study drug through end of treatment (~16 - 24 weeks)
  Phase 1b: Incidence and severity of treatment emergent adverse events (TEAEs)
Safety and tolerability | From first dose of study drug through end of treatment (~16 - 24 weeks)
  Phase Ia: Incidence and severity of treatment emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
The incidence of treatment emergent adverse events as assessed per CTCAE v5.0 | From first dose of study drug through end of study (~5 years)
  To assess safety and tolerability of [Ac-225]-PSMA-62
Time to initiation of any life-long ADT, or other systemic hormonal therapies for prostate cancer | From first dose of study drug through end of study (~5 years)
  OmHSPC only: Preliminary efficacy assessment
Absorbed dose estimates (Gy) in normal organs | From first dose of study drug through end of treatment (~16 - 24 weeks)
  Evaluation of the biodistribution and radiation dosimetry of [Ac-225]-PSMA-62 to normal organs
The proportion of patients with a PSA change from baseline | From first dose of study drug through efficacy follow-up period (up to approximately 3 years)
  To determine the effect of [Ac-225]-PSMA-62 on prostate-specific antigen (PSA) kinetics
Objective Response Rate (ORR) | From first dose of study drug until disease progression (up to approximately 3 years)
  mCRPC only: Percentage of participants with a complete response (CR) or partial response (PR)
Radiographic progression free survival (rPFS) | From first dose of study drug until disease progression (up to approximately 3 years)
  Phase Ib mCRPC only: rPFS per investigator assessment
Patient Reported Outcome (PRO) - Pain | From first dose of study drug until disease progression (up to approximately 3 years)
  Phase Ib only: Measured by the change on the Brief Pain Inventory Short Form (BPI-SF) questionnaire, scored from 0 ('No pain', 'Does not interfere') to 10 ('Pain as bad as you can imagine', 'Completely interferes') on the severity and interference on daily functions of pain.
Patient Reported Outcome (PRO) - Impact of treatment toxicity | From first dose of study drug until disease progression (up to approximately 3 years)
  Phase Ib only: Measured by the change the Functional Assessment of Cancer Therapy (FACT-Item GP5) questionnaire, scored from 0 ('Not at all') to 4 ('Very much') on the interference of symptoms related to treatment emergent adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- Canada (7):
  - Juravinski, Hamilton
  - Jewish General Hospital, Montreal
  - McGill University, Montreal
  - Centre Hospitalier Universite de QUEBEC, Québec
  - Hopital De Chicoutimi, Saguenay
  - Princess Margaret Cancer Centre, Toronto
  - BC Cancer Vancouver, Vancouver